CLINICAL TRIAL: NCT01801358
Title: A Phase Ib/II, Open-label, Multicenter Study of AEB071 and MEK162 in Adult Patients With Metastatic Uveal Melanoma
Brief Title: A Phase Ib/II Study of AEB071 and MEK162 in Adult Patients With Metastatic Uveal Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The trial was terminated for scientific reasons.
Sponsor: Array Biopharma, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Array BioPharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMEK162X2203
Record Dates: First submitted 2013-02-21; First posted 2013-02-28 (Estimated); Results first posted 2016-10-20 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Uveal Melanoma
Keywords: Melanoma,; melanoma of the eye,; uveal,; MEK162,; AEB071
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — sotrastaurin; binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): AEB071 and MEK162 combined
  Interventions: Drug: AEB071; Drug: MEK162
- Arm B (Experimental): MEK162 alone
  Interventions: Drug: MEK162

INTERVENTIONS:
Drug: AEB071 — Twice-daily doses of AEB071 for a cycle of 28-days, given without interruption (continuous cycles)
  Other Names: Sotrastaurin
  Arms: Arm A
Drug: MEK162 — Twice-daily doses of MEK162 for a cycle of 28-days, given without interruption (continuous cycles)

SUMMARY:
A phase Ib dose-escalation study of the AEB071 and MEK162 combination in adult patients with confirmed metastatic uveal melanoma. Cohorts of 3-6 patients will be assessed for dose limiting toxicities (DLTs) during Cycle 1 until the maximum tolerated dose (MTD) of the combination therapy is determined. The MTD or Phase 2 Recommended Dose (P2RD) will be used in a Phase II part of the study, which will enrol 55 patients each into two randomized groups: the combination therapy or MEK162 alone. The Phase II part will continue until proof of concept is established. Patients will continue treatment as long as clinical benefit is seen and no limiting adverse toxicity is observed

DETAILED DESCRIPTION:
Due to halted enrollment, the Phase II part of the study was not conducted. The Sponsor decided to permanently stop recruitment for the study prior to MTD determination.

Remaining patients on treatment with binimetinib and sotrastaurin who were considered by the Investigator to be benefiting from their treatment could have continued treatment and were to be followed up as per protocol. No patients were ongoing as of the data cut-off date. After the last patient last visit (LPLV) was declared, the study was terminated.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male and female patients aged 18 years or older
* A history of uveal (ocular) melanoma with biopsy-confirmed metastatic disease
* Consent to providing 3 tumor biopsy samples throughout the course of the study
* Presence of measurable disease
* A WHO performance status of less than or equal to 1

Exclusion Criteria:

* Presence of CNS lesions (stable lesions may be acceptable)
* Previous or concurrent malignancy, other than basal cell or squamous cell carcinoma of the skin: in situ carcinoma of the cervix, without evidence of recurrence for at least 3 years; a primary malignancy completely resected and no evidence of recurrence for at least 3 years
* Adverse event from prior chemotherapy, radiotherapy or surgery that has not recovered to CTCAE v4.03 Grade 1 or less, except for alopecia/sensory peripheral neuropathy, which must be less than Grade 2
* History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO
* Impaired cardiac function or clinically significant cardiac disease
* Impaired GI function or disease that could interfere with the absorption of AEB071 and/or MEK162
* Treatment with medicines or herbal supplements that are known inhibitors or inducers of CYP3A4/5 and cannot be withdrawn prior to study treatment
* Females of child-bearing potential who are unwilling or unable to use highly effective means of contraception
* Males who are unwilling or unable to use a condom during sexual intercourse
* Prior exposure to a MEK or PKC inhibitor Other inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (2):
  - Dana Farber Cancer Institute Dept. Onc, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center Dept of Onc.., New York, New York
- Pfizer Investigative Site, Paris, France
- Pfizer Investigative Site, Essen, Germany
- Pfizer Investigative Site, Leiden, Netherlands
- Pfizer Investigative Site, Madrid, Spain
- Pfizer Investigative Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The CMEK162X2203 study began recruitment on 26-Aug-2013 and concluded on 15-May-2015. Due to an enrollment halt, the Phase II part of the study was not conducted. The sponsor decided to permanently stop recruitment for the study prior to MTD determination.
Pre-assignment Details: Participant Flow and Baseline Demographics data represents the Full Analysis Set (FAS), which includes all patients who received at least one full or partial dose of sotrastaurin or binimetinib.
  Not completed subjects represents subjects that stopped treatment early, due to the corresponding reason.
Groups:
- Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (FAS); Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (FAS); Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (FAS); Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (FAS); Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (FAS); Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (FAS): Phase Ib (Dose Escalation)
  Phase Ib was the combination of sotrastaurin and binimetinib administered orally bid.
Period: Overall Study
Arm/Group | Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (FAS) | Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (FAS) | Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (FAS) | Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (FAS) | Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (FAS) | Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (FAS)
Started | 6 | 6 | 6 | 6 | 6 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 6 | 6 | 6 | 6 | 8
Not completed — Adverse Event | 0 | 2 | 1 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Progressive Disease | 6 | 4 | 4 | 5 | 6 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline Demographics data represents the Full Analysis Set (FAS), which includes all patients who received at least one full or partial dose of sotrastaurin or binimetinib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (FAS) | Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (FAS) | Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (FAS) | Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (FAS) | Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (FAS) | Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (FAS) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 5 | 3 | 4 | 5 | 27
  >=65 years | 1 | 1 | 1 | 3 | 2 | 3 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (15.21) | 57.0 (10.43) | 52.8 (10.82) | 59.8 (9.11) | 56.8 (10.87) | 61.5 (10.65) | 56.4 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 2 | 2 | 2 | 14
  Male | 3 | 4 | 3 | 4 | 4 | 6 | 24
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 1 | 1 | 2 | 1 | 1 | 0 | 6
  Russian | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown | 2 | 4 | 2 | 1 | 1 | 0 | 10
  Other | 2 | 1 | 2 | 4 | 4 | 8 | 21
Region of Enrollment [Number; unit: participants]
  Netherlands | 0 | 0 | 1 | 1 | 1 | 2 | 5
  United States | 1 | 0 | 2 | 2 | 2 | 0 | 7
  United Kingdom | 0 | 1 | 0 | 0 | 1 | 0 | 2
  France | 2 | 3 | 1 | 1 | 0 | 0 | 7
  Germany | 2 | 1 | 0 | 1 | 1 | 6 | 11
  Spain | 1 | 1 | 2 | 1 | 1 | 0 | 6
Baseline WHO Performance Status [Number; unit: participants] — Categories:
  * 0 - Fully active, able to carry on all pre-disease performance without restriction
  * 1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  * 2 - Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours
  * 3 - Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours
  * 4 - Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair
  participants
    0: | 3 | 6 | 5 | 5 | 5 | 8 | 32
    1: | 3 | 0 | 1 | 1 | 1 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Phase Ib: Incidence of Dose Limiting Toxicities (DLT) During the First Cycle
Description: A DLT is defined as an adverse event or abnormal laboratory value as defined in the protocol that is assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first 28 days of treatment with AEB071 and MEK162.
Time Frame: Cycle 1 (up to 28 days)
Population: Analysis is comprised of the Dose-determining Set, which is all patients from the safety set who either met the minimum exposure criterion below and had sufficient safety evaluations during Cycle 1, or discontinued earlier due to DLT during Cycle 1.
Measure: Number; unit: DLTs
Groups:
- Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (DDS); Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (DDS); Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (DDS); Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (DDS); Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (DDS); Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (DDS): Phase Ib (Dose Escalation)
  Phase Ib was the combination of sotrastaurin and binimetinib administered orally bid.
Arm/Group | Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (DDS) | Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (DDS) | Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (DDS) | Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (DDS) | Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (DDS) | Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (DDS)
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 4
DLTs
  Anaemia | 0 | 0 | 0 | 1 | 0 | 0
  Diarrhoea | 0 | 0 | 2 | 1 | 0 | 0
  Vomiting | 0 | 0 | 0 | 1 | 1 | 1
  Nausea | 0 | 0 | 0 | 1 | 0 | 1
  Fatigue | 0 | 0 | 1 | 1 | 0 | 0
  General Physical Health Deterioration | 0 | 0 | 1 | 0 | 0 | 0
  Malaise | 0 | 0 | 0 | 1 | 0 | 0
  Blood Creatinine Increased | 0 | 0 | 0 | 0 | 1 | 0
  Ejection Fraction Decreased | 0 | 0 | 0 | 0 | 0 | 1
  Dermatitis Acneiform | 0 | 2 | 0 | 0 | 0 | 0
  Rash | 0 | 0 | 0 | 1 | 0 | 0

2. Primary Outcome: Phase II: Progression Free Survival (PFS)
Description: The time from date of randomization to the date of event defined as the first documented progression or death due to any cause.
  Due to an enrollment halt, the Phase II part of the study was not conducted. The sponsor decided to permanently stop recruitment for the study prior to MTD determination.
Time Frame: From first dose of Cycle 1, Day 1 (C1D1) to time to progression (up to 18 months from Last Patient First Visit)
Groups:
- Phase II (Dose Expansion): Following the determination of the maximum tolerated dose (MTD) or the recommended phase two dose (RP2D), patients would have been randomized into two arms in a 1:1 ratio, to receive AEB071 and MEK162 or MEK162 alone. However, due to an enrollment halt, the Phase II part of the study did not occur.
Arm/Group | Phase II (Dose Expansion)
Number analyzed (Participants) | 0

3. Secondary Outcome: Phase Ib/II: The Number of Subjects Experiencing At Least One Adverse Event (AE)
Description: An adverse event is defined as the appearance of (or worsening of any pre-existing) undesirable sign(s), symptom(s), or medical condition(s) that occur after patient's signed informed consent has been obtained.
Time Frame: From first dose of Cycle 1, Day 1 (C1D1) to time to progression (up to 18 months from Last Patient First Visit)
Population: Analysis group consists of the Safety Set (SS), which is all patients who received at least one dose of AEB071 and MEK162, and have at least one valid post-baseline safety assessment.
Measure: Number; unit: participants
Groups:
- Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (SS); Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (SS); Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (SS); Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (SS); Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (SS); Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (SS): Phase Ib (Dose Escalation)
  Phase Ib was the combination of sotrastaurin and binimetinib administered orally bid.
Arm/Group | Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (SS) | Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (SS) | Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (SS) | Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (SS) | Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (SS) | Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (SS) | Phase II (Dose Expansion)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 0
participants | 6 | 6 | 6 | 6 | 6 | 8 |

4. Secondary Outcome: Phase Ib/II: The Number of Subjects Experiencing At Least One Serious Adverse Event (SAE)
Description: Serious adverse event (SAE) is defined as one of the following:
  * Is fatal or life-threatening
  * Results in persistent or significant disability/incapacity
  * Constitutes a congenital anomaly/birth defect
  * Is medically significant
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Note that hospitalizations for the following reasons should not be reported as serious adverse events:
    * Routine treatment or monitoring of the studied indication, not associated with any deterioration in condition
    * Elective or pre-planned treatment for a pre-existing condition that is unrelated to metastatic uveal melanoma and has not worsened since signing the informed consent
    * Social reasons and respite care in the absence of any deterioration in the patient's general condition
Time Frame: From first dose of Cycle 1, Day 1 (C1D1) to time to progression (up to 18 months from Last Patient First Visit)
Population: Analysis group is comprised of the Safety Set (SS), which is all patients who received at least one dose of AEB071 and MEK162, and have at least one valid post-baseline safety assessment.
Measure: Number; unit: participants
Arm/Group | Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (SS) | Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (SS) | Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (SS) | Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (SS) | Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (SS) | Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (SS) | Phase II (Dose Expansion)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8 | 0
participants | 3 | 1 | 3 | 4 | 2 | 6 |

5. Secondary Outcome: Phase Ib: Assessment of The Preliminary Anti-tumor Activity - Best Overall Response (BOR)
Description: Assessment of the preliminary anti-tumor activity of AEB071 and MEK162 in combination.
  The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for PD the smallest measurements recorded since the treatment started). In general, the patient's best response assignment will depend on the achievement of both measurement and confirmation criteria.
Time Frame: Cycle 1 (up to 28 days)
Population: Analysis group is comprised of the Full Analysis Set (FAS), which is all patients in the phase Ib part of the study who received at least one full or partial dose of AEB071 or MEK162.
Measure: Number; unit: participants
Arm/Group | Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (FAS) | Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (FAS) | Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (FAS) | Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (FAS) | Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (FAS) | Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (FAS)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8
participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 0 | 0
  Stable Disease | 5 | 4 | 4 | 2 | 3 | 5
  Progressive disease | 1 | 2 | 1 | 2 | 3 | 2
  Unknown | 0 | 0 | 1 | 2 | 0 | 1

6. Secondary Outcome: Phase Ib: Assessment of The Preliminary Anti-tumor Activity - Duration of Response (DOR)
Description: Assessment of the preliminary anti-tumor activity of AEB071 and MEK162 in combination.
  Duration of Response (DOR) is not reported, since there were no responses of Complete Response (CR) or Partial Response (PR) at any time during the study.
Time Frame: Cycle 1 (up to 28 days)
Population: as for outcome 5
Groups:
- Phase Ib (Dose Escalation): For Phase Ib, a minimum of three patients will be entered into each cohort and evaluated for safety (DLTs and any other medically significant event) at the end of Cycle 1.
  Phase Ib was the combination of sotrastaurin and binimetinib administered orally bid.
Arm/Group | Phase Ib (Dose Escalation)
Number analyzed (Participants) | 0

7. Secondary Outcome: Phase Ib: Assessment of The Preliminary Anti-tumor Activity - Progression Free Survival (PFS)
Description: Assessment of the preliminary anti-tumor activity of AEB071 and MEK162 in combination.
  PFS is the time from date of randomization/start of treatment to the date of event defined as the first documented progression or death due to any cause.
Time Frame: Cycle 1 (up to 28 days)
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (FAS) | Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (FAS) | Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (FAS) | Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (FAS) | Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (FAS) | Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (FAS)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 8
weeks | 3.6 [3.2 to 3.7] | 3.4 [1.6 to 3.7] | 4 [1.7 to 6.5] | 3.7 [1.2 to 5.3] | 3.1 [1.8 to 5.4] | 3.8 [1.9 to 11.5]

8. Secondary Outcome: Phase II: Evaluation of Preliminary Anti-tumor Activity - Overall Response Rate (CR+PR)
Description: Evaluation of the preliminary anti-tumor activity at the RP2D for AEB071 and MEK162 and at 45 mg BID for MEK162 alone.
  Overall response rate (ORR) is the proportion of patients with a best overall response of Complete Response (CR) or Partial Response (PR). This is also referred to as 'Objective response rate' in some protocols or publications.
  Due to an enrollment halt, the Phase II part of the study was not conducted.
Time Frame: From first dose of Cycle 1, Day 1 (C1D1) to time to progression (up to 18 months from Last Patient First Visit)
Population: as for outcome 5
Arm/Group | Phase II (Dose Expansion)
Number analyzed (Participants) | 0

9. Secondary Outcome: Phase II: Evaluation of Preliminary Anti-tumor Activity - Best Overall Response (BOR)
Description: Evaluation of the preliminary anti-tumor activity at the RP2D for AEB071 and MEK162 and at 45 mg BID for MEK162 alone.
  The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for Progressive Disease (PD) the smallest measurements recorded since the treatment started). In general, the patient's best response assignment will depend on the achievement of both measurement and confirmation criteria.
  Due to an enrollment halt, the Phase II part of the study was not conducted.
Time Frame: From first dose of Cycle 1, Day 1 (C1D1) to time to progression (up to 18 months from Last Patient First Visit)
Population: as for outcome 5
Arm/Group | Phase II (Dose Expansion)
Number analyzed (Participants) | 0

10. Secondary Outcome: Phase II: Evaluation of Preliminary Anti-tumor Activity - Duration of Response (DOR)
Description: Evaluation of the preliminary anti-tumor activity at the RP2D for AEB071 and MEK162 and at 45 mg BID for MEK162 alone.
  Duration of Response is not reported, due to the enrollment halt, which occurred prior to Phase II of the study.
Time Frame: From first dose of Cycle 1, Day 1 (C1D1) to time to progression (up to 18 months from Last Patient First Visit)
Population: as for outcome 5
Arm/Group | Phase II (Dose Expansion)
Number analyzed (Participants) | 0

11. Secondary Outcome: Phase II: Evaluation of Preliminary Anti-tumor Activity - Overall Survival (OS)
Description: Evaluation of the preliminary anti-tumor activity at the RP2D for AEB071 and MEK162 and at 45 mg BID for MEK162 alone.
  Overall survival (OS) is defined as the time from date of randomization/start of treatment to date of death due to any cause.
  Due to an enrollment halt, the Phase II part of the study was not conducted.
Time Frame: From first dose of Cycle 1, Day 1 (C1D1) to time to progression (up to 18 months from Last Patient First Visit)
Population: as for outcome 5
Arm/Group | Phase II (Dose Expansion)
Number analyzed (Participants) | 0

12. Secondary Outcome: Phase Ib: PK Parameters for AEB071 - AUC0-8hr (Cycle 1; Day 1)
Description: Blood samples were collected from all patients during Cycle 1 (Days 1 and 15) for pharmacokinetic profiling. On Days 8 and 22 of Cycle 1, trough samples were collected. Additionally, pre-dose samples were collected on Day 1 of Cycle 2 through Cycle 6.
Time Frame: Cycle 1 (Day 1)
Population: This analysis group is comprised of the Pharmacokinetic Analysis Set (PAS), which is all patients who have evaluable pharmacokinetic (PK) data. The PAS will be used for summaries (tables and figures) and listings of PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/ml
Groups:
- Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (PAS); Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (PAS); Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (PAS); Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (PAS); Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (PAS); Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (PAS): Phase Ib (Dose Escalation)
  Phase Ib was the combination of sotrastaurin and binimetinib administered orally bid.
Arm/Group | Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (PAS) | Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (PAS) | Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (PAS)
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 4 | 8
hr*ng/ml | 7448.5 (46.34) | 7136 (25.09) | 15090 (53.89) | 14051.2 (45.83) | 18840.8 (36.24) | 15217.1 (71.48)

13. Secondary Outcome: Phase lb: PK Parameters for AEB071 - Cmax (Cycle 1; Day 1)
Description: as for outcome 12
Time Frame: Cycle 1 (Day 1)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (PAS) | Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (PAS) | Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (PAS)
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 4 | 8
ng/ml | 1837.5 (35.9) | 1932.5 (31.18) | 2968.1 (58.32) | 2813 (36.83) | 4459 (26.45) | 3768.7 (57.12)

14. Secondary Outcome: Phase lb: PK Parameters for AEB071 - Tmax (Cycle 1; Day 1)
Description: as for outcome 12
Time Frame: Cycle 1 (Day 1)
Population: as for outcome 12
Measure: Median (Full Range); unit: hr
Arm/Group | Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (PAS) | Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (PAS) | Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (PAS)
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 4 | 8
hr | 1.6 [0.4 to 4] | 1.1 [1 to 4] | 1.5 [0.5 to 2] | 1 [0.5 to 1.9] | 1 [1 to 2] | 2.1 [0.5 to 5.8]

15. Secondary Outcome: Phase Ib: PK Parameters for AEB071 - AUC0-8hr (Cycle 1; Day 15)
Description: as for outcome 12
Time Frame: Cycle 1 (Day 15)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/ml
Arm/Group | Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (PAS) | Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (PAS) | Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (PAS)
Number analyzed (Participants) | 6 | 4 | 2 | 5 | 5 | 5
hr*ng/ml | 5879.9 (32.46) | 6330.3 (29.28) | 16737.1 (17.56) | 15313.6 (105.21) | 15055.5 (78.89) | 20629.7 (11.81)

16. Secondary Outcome: Phase lb: PK Parameters for AEB071 - Cmax (Cycle 1; Day 15)
Description: as for outcome 12
Time Frame: Cycle 1 (Day 15)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (PAS) | Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (PAS) | Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (PAS)
Number analyzed (Participants) | 6 | 4 | 2 | 5 | 5 | 5
ng/ml | 1244.6 (27.5) | 1347.1 (28.56) | 3065.6 (60.1) | 3263.8 (96.11) | 3597.2 (62.84) | 3716.5 (23.72)

17. Secondary Outcome: Phase lb: PK Parameters for AEB071 - Tmax (Cycle 1; Day 15)
Description: as for outcome 12
Time Frame: Cycle 1 (Day 15)
Population: as for outcome 12
Measure: Median (Full Range); unit: hr
Arm/Group | Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (PAS) | Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (PAS) | Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (PAS)
Number analyzed (Participants) | 6 | 4 | 2 | 5 | 5 | 5
hr | 2 [1.1 to 8.3] | 1.5 [0.5 to 2] | 2.6 [1 to 4.2] | 3.9 [2 to 4.2] | 1.9 [0.5 to 2.1] | 2.1 [2 to 8]

18. Secondary Outcome: Phase Ib: PK Parameters for MEK162 - AUC0-8hr (Cycle 1; Day 1)
Description: as for outcome 12
Time Frame: Cycle 1 (Day 1)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/ml
Arm/Group | Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (PAS) | Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (PAS) | Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (PAS)
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 5 | 8
hr*ng/ml | 1587.7 (55.75) | 1496.7 (30.02) | 1088.7 (49.45) | 1590.5 (43.49) | 984.4 (72.57) | 962 (50.15)

19. Secondary Outcome: Phase lb: PK Parameters for MEK162 - Cmax (Cycle 1; Day 1)
Description: as for outcome 12
Time Frame: Cycle 1 (Day 1)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (PAS) | Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (PAS) | Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (PAS)
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 5 | 8
ng/ml | 362 (46.74) | 432.6 (56.3) | 245.4 (63.08) | 328.4 (59.07) | 243.5 (53.27) | 222.8 (58.13)

20. Secondary Outcome: Phase lb: PK Parameters for MEK162 - Tmax (Cycle 1; Day 1)
Description: as for outcome 12
Time Frame: Cycle 1 (Day 1)
Population: as for outcome 12
Measure: Median (Full Range); unit: hr
Arm/Group | Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (PAS) | Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (PAS) | Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (PAS)
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 5 | 8
hr | 1.1 [1 to 3.8] | 1.1 [1 to 4.1] | 2 [1 to 2.1] | 4 [0.5 to 4.1] | 2 [0.6 to 2.3] | 1.1 [0.5 to 4]

21. Secondary Outcome: Phase Ib: PK Parameters for MEK162 - AUC0-8hr (Cycle 1; Day 15)
Description: as for outcome 12
Time Frame: Cycle 1 (Day 15)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/ml
Arm/Group | Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (PAS) | Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (PAS) | Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (PAS)
Number analyzed (Participants) | 6 | 4 | 4 | 4 | 5 | 4
hr*ng/ml | 1807.4 (43.6) | 1927.9 (42.48) | 1374.2 (68.21) | 1454.7 (41.13) | 1268.5 (70.41) | 1275.8 (39.04)

22. Secondary Outcome: Phase lb: PK Parameters for MEK162 - Cmax (Cycle 1; Day 15)
Description: as for outcome 12
Time Frame: Cycle 1 (Day 15)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (PAS) | Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (PAS) | Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (PAS)
Number analyzed (Participants) | 6 | 4 | 4 | 4 | 5 | 4
ng/ml | 454.5 (42.42) | 418.9 (34.62) | 307 (88.45) | 362.7 (59.8) | 340.7 (80.64) | 284.1 (52.79)

23. Secondary Outcome: Phase lb: PK Parameters for MEK162 - Tmax (Cycle 1; Day 15)
Description: as for outcome 12
Time Frame: Cycle 1 (Day 15)
Population: as for outcome 12
Measure: Median (Full Range); unit: hr
Arm/Group | Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (PAS) | Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (PAS) | Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (PAS) | Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (PAS)
Number analyzed (Participants) | 6 | 4 | 4 | 4 | 5 | 4
hr | 2 [1.1 to 8.3] | 1.6 [1.1 to 4] | 3 [1 to 8.2] | 2.9 [2 to 4.1] | 1.9 [0.5 to 2.1] | 1.5 [0.5 to 8]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected for approximately 2 years (August, 2013 through May, 2015), which was the duration of the trial.
Description: AE reporting is comprised of the Safety Set (SS), which is all patients who received at least one dose of AEB071 and MEK162, and have at least one valid post-baseline safety assessment.
Arm/Group | Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (SS) | Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (SS) | Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (SS) | Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (SS) | Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (SS) | Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (SS)
Serious Adverse Events (participants affected / at risk) | 3/6 | 1/6 | 3/6 | 4/6 | 2/6 | 6/8
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 6/6 | 6/6 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (SS) (N=6) | Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (SS) (N=6) | Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (SS) (N=6) | Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (SS) (N=6) | Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (SS) (N=6) | Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (SS) (N=8)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALAISE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ASCITES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATOMEGALY (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase Ib: AEB071 150 mg Bid + MEK162 45 mg Bid (SS) (N=6) | Phase Ib: AEB071 200 mg Bid + MEK162 45 mg Bid (SS) (N=6) | Phase Ib: AEB071 300 mg Bid + MEK162 30 mg Bid (SS) (N=6) | Phase Ib: AEB071 300 mg Bid + MEK162 45 mg Bid (SS) (N=6) | Phase Ib: AEB071 350 mg Bid + MEK162 30 mg Bid (SS) (N=6) | Phase Ib: AEB071 400 mg Bid + MEK162 30 mg Bid (SS) (N=8)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 3 (3) | 4 (4) | 3 (3) | 3 (3) | 3 (3) | 5 (5)
OEDEMA PERIPHERAL (General disorders) | 2 (2) | 2 (2) | 4 (4) | 3 (3) | 2 (2) | 3 (3)
ASTHENIA (General disorders) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 3 (3)
PYREXIA (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MALAISE (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
CHILLS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 4 (4) | 5 (5) | 1 (1) | 2 (2) | 3 (3) | 2 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 4 (4) | 1 (1) | 3 (3) | 3 (3) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 2 (2)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EJECTION FRACTION DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WEIGHT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
CEREBROVASCULAR DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHORIORETINOPATHY (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
RETINAL DETACHMENT (Eye disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
VISUAL IMPAIRMENT (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
CATARACT (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EYE DISORDER (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EYELID OEDEMA (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MACULAR OEDEMA (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
PERIORBITAL OEDEMA (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
RETINAL OEDEMA (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RETINOPATHY (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 6 (6) | 5 (5) | 6 (6) | 6 (6) | 6 (6) | 8 (8)
NAUSEA (Gastrointestinal disorders) | 6 (6) | 3 (3) | 4 (4) | 6 (6) | 4 (4) | 7 (7)
VOMITING (Gastrointestinal disorders) | 5 (5) | 3 (3) | 5 (5) | 5 (5) | 5 (5) | 7 (7)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEPATIC PAIN (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHROMATURIA (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
RENAL COLIC (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
RASH (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 1 (1)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 3 (3) | 3 (3) | 2 (2) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH FOLLICULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
XERODERMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
CACHEXIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RASH PUSTULAR (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2)

LIMITATIONS AND CAVEATS:
Due to an enrollment halt, the Phase II part of the study was not conducted. The sponsor decided to permanently stop recruitment for the study prior to MTD determination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of the sponsor's agreements with its investigators may vary. However, the sponsor does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e. data from all sites) in the clinical trial.